CLINICAL TRIAL: NCT03175003
Title: Assessment of Protein Intake and Micronutrient Fortification in Metabolically at Risk Children
Brief Title: Assessment of a New Food Product in Metabolically at Risk Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1009239
Record Dates: First submitted 2017-02-13; First posted 2017-06-05 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Risk Factor; Inflammation; Micronutrient Deficiency
MeSH Terms: conditions — Inflammation | interventions — Food

STUDY DESIGN:
Intervention Model Description: Double blind, controlled, 4 parallel arm design
Who Masked: Participant, Investigator
Masking Description: Products will look and taste similar, and will be provided in coded packaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Food Product 1 (Active Comparator): Macronutrient similar to experimental, micronutrient lower than experimental
  Interventions: Other: Food Product
- Food Product 2 (Active Comparator): Macronutrient lower than experimental, micronutrient similar to experimental
  Interventions: Other: Food Product
- Food Product 3 (Experimental): Experimental 1
  Interventions: Other: Food Product
- Food Product 4 (Experimental): Experimental 2
  Interventions: Other: Food Product

INTERVENTIONS:
Other: Food Product — Each food product will provide similar calories, but a different micro- and macro-nutrient composition

SUMMARY:
The current study conducted will lend toward the optimization of the development of a food product that will promote a shift towards improved metabolic health. Specifically, this trial will determine the optimal level of protein needed to elicit positive changes in markers of inflammation, metabolic and micronutrient status, hepatic lipid metabolism, vascular function, and the relationship of these changes to the metabolome in school aged children (9 - 13 years of age).

DETAILED DESCRIPTION:
Each participant will be asked to participate in a screening and 2 study intervention visits. Each intervention visit will include anthropometric measures, complete the education component, vascular function tests, and a blood draw and spot urine. The screening visit will confirm the child's eligibility for study enrollment and will serve to acclimate the child to the vascular function, and physical activity measurements. The remaining 2 visits will be scheduled 4 weeks apart. The participants will also be provided and asked to wear a physical activity monitor, which in addition to tracking physical activity, will also be used to incorporate a nutrition education program. The parent/guardian will be asked to help with providing the child the daily food product and to help their child fill out the compliance log. Volunteers will also be sought for stool and saliva collection.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 9-13 years old
* Subject is willing and able to comply with the study protocols
* Subject is willing to consume the test products
* Access to a smart phone or tablet at least 1x / week; and willing to download a free applications associated with the study

Exclusion Criteria:

* Allergies or intolerances to peas, legumes, pulses, soy, dairy or wheat/gluten
* Under current medical supervision
* Tanner Score = 4
* Non-English speaking
* Current participation in a daily exercise routine of moderate or high intensity
* Self-reported presence of disease, a history of serious illness, or who are currently under acute medical care.
* Currently taking prescription drugs or supplements
* Any supplement use, including multi-vitamin/ mineral, herbal, plant or botanical, fish oil, and oil supplements.
* Self-reported malabsorption or gastrointestinal issues
* Current enrollee in a clinical research study.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Microvascular Function | Compare change in baseline and 4 weeks
  Measured by EndoPAT2000. A PAT (Peripheral Arterial Tone) ratio is created using the post and pre occlusion values

SECONDARY OUTCOMES:
Change in Metabolome | Compare change in baseline and 4 weeks
  Measured with Nuclear Magnetic Resonance (NMR)
Change in Lipidome | Compare change in baseline and 4 weeks
  Measured by Ultra Performance Liquid Chromatography (UPLC) tandem mass-spectrometry
Change in Inflammatory Markers | Compare change in baseline and 4 weeks
  Measured by immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No